CLINICAL TRIAL: NCT06716437
Title: Digitally Enabled Prehabilitation in a Community-based Setting for Patients Undergoing Lung Cancer Surgery
Brief Title: Prehabilitation for Patients Undergoing Lung Cancer Surgery
Acronym: DIGI-Lung
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); St Vincent's Hospital Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30930
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Prehabilitation; Inspiratory Muscle Training; Exercise Therapy; Lung Cancer; Telehealth
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prehabilitation arm (Experimental): Patients will receive the prehabilitation program
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Patients will undergo a physiotherapy-led digitally-enabled prehabilitation program before lung resection surgery.
  The intervention will be delivered through a mobile app and supported by tele-health and will consist of:
  i) watching six educational videos embedded on the app on relevant topics to prepare for surgery, such as the importance of physical fitness, breathing exercises after surgery, and pain management.
  ii) a physical activity coaching program to increase daily activity with feedback iii) a home-based, unsupervised exercise program consisting of 10 whole body strengthening exercises delivered in a video format iv) an inspiratory muscle training program using a hand-held device to be performed twice daily.

SUMMARY:
Major surgery has been linked to running a marathon as in both represent large endeavours where the body will experience an increase in demands to supply the necessary energy. It has been alledged that, as one would train to prepare for a marathon, the same should be applied to surgery. The process of getting ready and/or fitter for surgery is frequently referred to as prehabilitation and it usually involves interventions on improving nutrition and diet, getting fit and improve emotional wellness. Prehabilitation can improve the recovery after surgery and reduce the time spent in hospital afterwards. This research seeks to determine whether a home based program of increased physical activity and breathing training can improve patients' physical and respiratory function in preparation for lung cancer surgery.

DETAILED DESCRIPTION:
Patients with lung cancer who are scheduled to undergo lung resection surgery will be provided with a digitally-enabled, remotely-monitored prehablitation program. The intervention will consist of the following components: i) general education; ii) inspiratory muscle training; iii) physical activity coaching; and iv) home-based exercise training. The program will be supported with a mobile app and weekly telehealth sessions with one experienced physiotherapist. Participants will be assessed at baseline and at the end of the intervention, prior to surgery. Participants will be contacted and scheduled to undergo face-to-face assessments on lung function, respiratory muscle strength, and functional capacity both at baseline and after the prehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer and scheduled for lung resection surgery
* Ability to understand and speak English to follow instructions and complete the intended assessments.
* Age ≥ 18 years at the point of baseline screening
* Provide written informed consent for the trial
* Sufficient digital literacy to use a smartphone and mobile app
* No contraindications for exercise

Exclusion Criteria:

* Other cancer diagnoses than lung cancer
* Surgery scheduled in less than one week
* Unstable psychiatric, cognitive or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | From enrollment to the end of the study approximately one week after surgery
  Feasibility of the intervention determined by enrolment rate (number of patients who accept participation in the trial vs. number of eligible patients)
App usability and acceptability | Within one week before surgery
  The app usability will be measured with a questionnaire (the mHealth App Usability Questionnaire). The questionnaire consists of 21 items on a likert scale ranging from 1 (disagree) to 7 (agree) assessing different domains of a mHealth app. A median of 4.5 out of 7 across all domains will be considered as high usability and acceptability.

SECONDARY OUTCOMES:
Safety of the intervention | From enrollment to the end of the program before surgery
  Adverse events, defined as any unexpected, undesirable event, such as injury, fall, and discomfort related to prehabilitation program will be recorded weekly through telehealth. They will be classified according to the Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.
Inspiratory Muscle Strength | Within one week before surgery
  Maximal inspiratory pressure (MIP) registered at the mouth will be recorded using a specific device (BHC RP Check, Bird Health Care Australia).
Diaphragmatic excursion and thickness | Within one week before surgery
  Diaphragmatic excurssion will be measured with through Point of Care Ultrasound (POCUS) both at normal breathing and maximal inspiration. Diaphragmatic thickness will also be measured.
Lung function | Within one week before surgery
  Lung function parameters including forced vital capacity (FVC) and forced expiratory volume in the first second (FEV1) will be collected during a forced spirometry test. The tests will be conducted according to the international recommendations from the ATS/ERS.
Self-efficacy | Within one week before surgery
  Patient's perception of self-efficacy will be measured using a validated questionnaire (General Self-Efficacy Scale). The scale is 10-item each one measured on a likert-scale from 1 to 4. Total scores range from 10 to 40 with higher scores indicating higher self-efficacy.
Participant satisfaction | Within one week before surgery
  Participants' satisfaction with the intervention will be measured through the Australian Hospital Patient Experience Question Set (AHPEQS). The AHPEQS is a 12-item questionnaire with each question assessed on a likert-scale which measures the satisfaction with a healthcare intervention. There is no scoring for this scale.
Health Related Quality of Life | Within one week before surgery
  Heaht-related quality of life will be assessed using a validated questionnaire specific to cancer patients from the European Organization of Research in Cancer Treatment (EORTC QLQ C30). The questionnaire will be self-administered and consists of 30 questions on several domains of physical functioning, emotional functioning and cancer-related symptoms. Two main subscales are obtained from the questionnaire (one in function, one in symptoms) plus one item on global health. The score ranges from 0 to 100 with higher scores representing higher self-reported quality of life or higher symptom burden.
Recovery from surgery | Within one week before surgery
  Self-reported recovery from surgery will be measured using a validated questionnaire (the Quality of Recovery Questionnaire - QoR15).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Denehy, PhD, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Department of Physiotherapy, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be considered upon reasonable request made to the principal investigator

REFERENCES:
- [Background] Waterland JL, Ismail H, Amin B, Granger CL, Denehy L, Riedel B. Patient acceptance of prehabilitation for major surgery: an exploratory survey. Support Care Cancer. 2021 Feb;29(2):779-785. doi: 10.1007/s00520-020-05547-1. Epub 2020 May 28. PMID 32462351
- [Background] Whish-Wilson GA, Edbrooke L, Cavalheri V, Denehy L, Seller D, Granger CL, Parry SM. Physiotherapy and Exercise Management of People Undergoing Surgery for Lung Cancer: A Survey of Current Practice across Australia and New Zealand. J Clin Med. 2023 Mar 9;12(6):2146. doi: 10.3390/jcm12062146. PMID 36983146
- [Background] Kunadharaju R, Saradna A, Ray A, Yu H, Ji W, Zafron M, Mador MJ. Post-Operative Outcomes of Pre-Thoracic Surgery Respiratory Muscle Training vs Aerobic Exercise Training: A Systematic Review and Network Meta-analysis. Arch Phys Med Rehabil. 2023 May;104(5):790-798. doi: 10.1016/j.apmr.2022.10.015. Epub 2022 Dec 17. PMID 36539175
- [Background] Ferreira V, Lawson C, Ekmekjian T, Carli F, Scheede-Bergdahl C, Chevalier S. Effects of preoperative nutrition and multimodal prehabilitation on functional capacity and postoperative complications in surgical lung cancer patients: a systematic review. Support Care Cancer. 2021 Oct;29(10):5597-5610. doi: 10.1007/s00520-021-06161-5. Epub 2021 Mar 25. PMID 33768372
- [Background] Sebio Garcia R, Yanez Brage MI, Gimenez Moolhuyzen E, Granger CL, Denehy L. Functional and postoperative outcomes after preoperative exercise training in patients with lung cancer: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):486-97. doi: 10.1093/icvts/ivw152. Epub 2016 May 25. PMID 27226400
- [Background] Cavalheri V, Granger CL. Exercise training as part of lung cancer therapy. Respirology. 2020 Nov;25 Suppl 2:80-87. doi: 10.1111/resp.13869. Epub 2020 Jun 1. PMID 32567236
- [Background] Cavalheri V, Granger C. Preoperative exercise training for patients with non-small cell lung cancer. Cochrane Database Syst Rev. 2017 Jun 7;6(6):CD012020. doi: 10.1002/14651858.CD012020.pub2. PMID 28589547